CLINICAL TRIAL: NCT01292291
Title: PROMIS - Prostate MRI Imaging Study - Evaluation of Multi-Parametric Magnetic Resonance Imaging in the Diagnosis and Characterization of Prostate Cancer
Brief Title: MRI in Diagnosing Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College London Hospitals (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: MRC-PR11; CDR0000694647 (Registry Identifier: PDQ (Physician Data Query)); EU-21104; UCL-11/009; ISRCTN16082556 (Registry Identifier: ISRCTN (International Standard Randomised Controlled Trial Number Register))
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2011-09

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIA prostate cancer; stage IIB prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Other: biologic sample preservation procedure
Other: laboratory biomarker analysis
Other: study of socioeconomic and demographic variables
Procedure: diffusion-weighted magnetic resonance imaging
Procedure: dynamic contrast-enhanced magnetic resonance imaging
Procedure: multiparametric magnetic resonance imaging
Procedure: quality-of-life assessment
Procedure: transperineal prostate biopsy
Procedure: transrectal prostate biopsy
Procedure: ultrasound-guided prostate biopsy

SUMMARY:
RATIONALE: Diagnostic procedures, such as magnetic resonance imaging (MRI), may help find prostate cancer and learn the extent of disease.

PURPOSE: This clinical trial is studying the safety of MRI and to see how well it works in diagnosing prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the ability of multiparametric magnetic resonance imaging (MP-MRI) to identify men who can safely avoid unnecessary biopsy.
* To assess the ability of the MP-MRI-based diagnostic pathway to improve the rate of detection of clinically significant cancer as compared to transrectal ultrasound (TRUS) biopsy.
* To estimate the cost-effectiveness of an MP-MRI based diagnostic pathway.

OUTLINE: This is a multicenter study.

Patients undergo multiparametric magnetic resonance imaging (MRI) (T2-weighted imaging, diffusion-weighted MRI, and dynamic contrast-enhanced MRI) followed by template prostate mapping and transrectal ultrasound biopsy.

Some patients may undergo blood, urine, and tissue sample collection periodically for biomarker studies. Samples are banked for future research analysis.

Patients complete a quality-of-life questionnaire (EQ-5D) at baseline, during, and after completion of study. An economic analysis will be performed for cost-effectiveness.

After completion of study intervention, patients are followed up periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Men at risk of prostate cancer who have been advised to have a prostate biopsy
* Suspected stage ≤ T2 on rectal examination (organ confined)
* Serum PSA ≤ 15 ng/mL within the past 3 months

PATIENT CHARACTERISTICS:

* Fit for general/spinal anesthesia
* Fit to undergo all protocol procedures including a transrectal ultrasound
* No evidence of a urinary tract infection or history of acute prostatitis within the past 3 months
* No contraindication to MRI (e.g., claustrophobia, pacemaker, or estimated GFR ≤ 50)
* No other medical condition precluding procedures described in the protocol

PRIOR CONCURRENT THERAPY:

* No prior prostate biopsy, prostate surgery, or treatment for prostate cancer (interventions for benign prostatic hyperplasia/bladder outflow obstruction are acceptable)
* No prior hip replacement surgery

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 714 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Safety of multiparametric magnetic resonance imaging (MP-MRI)
Recruitment
Proportion of men who could safely avoid biopsy as determined by specificity and negative predictive values
Proportion of men correctly identified by MP-MRI to have clinically significant prostate cancer as determined by sensitivity and positive predictive values

SECONDARY OUTCOMES:
Proportion of men who could safely avoid biopsy
Proportion of men testing positive on MP-MRI
Performance characteristics of TRUS versus template prostate mapping (TPM)
Evaluation of the optimal combination of MP-MRI functional parameters
Intra-observer variability in the reporting of MP-MRI
Evaluation of socio-demographic, clinical, imaging and radiological variables in relation to the detection of clinically significant prostate cancer
Health-related quality of life using the EQ-5D questionnaire
Resource use and costs for further economic evaluation
Translational research

CONTACTS AND LOCATIONS:
Overall Officials: Mark Emberton, MD, FRCS, MBBS, Principal Investigator — University College London Hospitals

REFERENCES:
- [Derived] Stavrinides V, Norris JM, Karapanagiotis S, Giganti F, Grey A, Trahearn N, Freeman A, Haider A, Carmona Echeverria LM, Bott SRJ, Brown LC, Burns-Cox N, Dudderidge TJ, El-Shater Bosaily A, Ghei M, Henderson A, Hindley RG, Kaplan RS, Oldroyd R, Parker C, Persad R, Rosario DJ, Shergill IS, Winkler M, Kirkham A, Punwani S, Whitaker HC, Ahmed HU, Emberton M; PROMIS Group. Regional Histopathology and Prostate MRI Positivity: A Secondary Analysis of the PROMIS Trial. Radiology. 2023 Apr;307(1):e220762. doi: 10.1148/radiol.220762. Epub 2022 Dec 13. PMID 36511804
- [Derived] Brown LC, Ahmed HU, Faria R, El-Shater Bosaily A, Gabe R, Kaplan RS, Parmar M, Collaco-Moraes Y, Ward K, Hindley RG, Freeman A, Kirkham A, Oldroyd R, Parker C, Bott S, Burns-Cox N, Dudderidge T, Ghei M, Henderson A, Persad R, Rosario DJ, Shergill I, Winkler M, Soares M, Spackman E, Sculpher M, Emberton M. Multiparametric MRI to improve detection of prostate cancer compared with transrectal ultrasound-guided prostate biopsy alone: the PROMIS study. Health Technol Assess. 2018 Jul;22(39):1-176. doi: 10.3310/hta22390. PMID 30040065
- [Derived] Ahmed HU, El-Shater Bosaily A, Brown LC, Gabe R, Kaplan R, Parmar MK, Collaco-Moraes Y, Ward K, Hindley RG, Freeman A, Kirkham AP, Oldroyd R, Parker C, Emberton M; PROMIS study group. Diagnostic accuracy of multi-parametric MRI and TRUS biopsy in prostate cancer (PROMIS): a paired validating confirmatory study. Lancet. 2017 Feb 25;389(10071):815-822. doi: 10.1016/S0140-6736(16)32401-1. Epub 2017 Jan 20. PMID 28110982